CLINICAL TRIAL: NCT07297628
Title: The Effect of the '1 Concept-1 Minute' Game on the Perception of Caring in Teaching Care: A Randomized Controlled Study
Brief Title: Teaching Caring Through '1 Concept-1 Minute
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUS-HEM-CO-04
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Student
Keywords: '1 Concept-1 Minute' Game; Teaching Care

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized controlled interventional trial. Participants were randomly assigned to two groups: the intervention group, which received game-based learning via the "One Concept-One Minute" method, and the control group, which continued with traditional lecture-based instruction. The aim of the study is to evaluate the effectiveness of the game-based approach on nursing students' concept comprehension and learning motivation within the scope of a health assessment course.
Masking Description: Investigators were blinded to group assignment (intervention or control) to reduce potential bias in data collection and interpretation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants in the control group will receive traditional lecture-based instruction on nursing care behaviors, without the use of any game-based or interactive strategies.
- Experimental Arm (Experimental): In this group, the "1 Concept-1 Minute" game-based learning method will be applied at the end of the "Care Behaviors" course over a period of two weeks, totaling 4 hours. At the end of each session, students will randomly select a care-related concept covered in the course and explain it to their classmates within one minute. This intervention is designed to promote active participation, strengthen the understanding of nursing care concepts, and enhance student motivation through a fun and interactive educational approach.
  Interventions: Behavioral: 1 Concept-1 Minute Game-Based Learning Method

INTERVENTIONS:
Behavioral: 1 Concept-1 Minute Game-Based Learning Method — This intervention is a game-based learning activity titled "1 Concept-1 Minute," designed for nursing students. At the end of each class session, students randomly select one care-related concept and are given one minute to explain it to their peers. The activity will be implemented over two weeks, with two sessions lasting two hours each (total 4 hours). The goal of the intervention is to reinforce students' understanding of care-related concepts, enhance their communication skills, and increase motivation through active learning.
  Other Names: Experimental Arm
  Arms: Experimental Arm

SUMMARY:
This study aims to evaluate the effectiveness of a gamified learning strategy called "1 Concept-1 Minute" on nursing students' understanding of care concepts and their learning motivation. Conducted within the context of a Health Assessment course in a nursing education program, this quasi-experimental research investigates whether game-based learning methods enhance students' cognitive engagement and comprehension in clinical education. Given the global need for competent nursing professionals and the limitations in clinical placements, innovative, student-centered approaches such as this game are crucial to improving learning outcomes. The study is based on the Self-Determination Theory (SDT) framework to interpret motivational impacts.

DETAILED DESCRIPTION:
Knowledge and practice training is a fundamental component of healthcare courses. In this context, instructors are expected to foster professional thinking skills that support learning and exploration among students, provide opportunities to apply acquired knowledge, and equip them with the knowledge, skills, and attitudes necessary to manage various clinical situations. Within nursing programs, the Health Assessment course is a compulsory subject that focuses on collecting health data from patients to identify potential health problems. Therefore, in addition to learning normal and abnormal health conditions, students must also adequately understand prerequisite topics such as care and treatment in order to perform health assessments correctly.

Clinical education is a critical component of nursing training, integrating theoretical knowledge with practical skills. However, previous studies have highlighted various factors that negatively affect the acquisition of clinical competencies. These include limited clinical placement opportunities despite increasing student numbers, a shortage of nursing educators, student stress, insufficient integration of theory and practice, and the resulting anxiety and frustration.

Effective strategies are required to address the global nursing shortage, prevent academic underperformance, and enhance professional competence. Recent research has shown that gamification and serious games have the potential to improve the quality of healthcare professional education. Integrating game-based learning strategies can increase motivation and engagement. However, the exact impact of such approaches on nursing students remains unclear. This highlights the importance of the current study and the need for further research.

In this context, our study aims to identify, evaluate, and summarize the effectiveness of game-based approaches in nursing education in terms of student learning outcomes and perceptions. Although game-based learning plays a significant role in increasing motivation and engagement, the lack of a unified theory of gamification means that this research is not based on a specific theoretical framework. However, the Self-Determination Theory (SDT) is acknowledged to play a critical role in game design and gamified learning experiences.

A review of the literature reveals a limited number of studies focusing on the use of short, effective, and student-centered methods for teaching care concepts in nursing education. The aim of this study is to examine the effect of the "1 Concept-1 Minute" game on nursing students' understanding of care concepts and their learning motivation.

ELIGIBILITY:
Inclusion Criteria:

* Willing to continue their education throughout the study period, Voluntarily agreeing to participate in the study and signing the informed consent form,

Exclusion Criteria:

* Having previously participated in a similar game-based learning or "1 Concept 1 Minute" training, Having health conditions or other reasons preventing attendance during the study period, Students unwilling to continue participation or who do not provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Care Behavior Scale-30 Score | Measured immediately after the 2-week intervention period (4 hours total)
  The Care Behavior Scale-30, a validated instrument assessing nursing care perceptions and behaviors, will be used to evaluate changes in participants' nursing care attitudes and behaviors before and after the intervention. The scale consists of 30 items scored on a 6-point Likert scale, with total scores ranging from 30 to 180. Higher scores indicate better care behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Faculty of Nursing, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We do not plan to share Individual Participant Data (IPD) due to concerns regarding participant confidentiality and the need to protect their privacy.